CLINICAL TRIAL: NCT00680953
Title: A Randomized, Double-Blind, Placebo-controlled Phase 3 Study Evaluating Efficacy and Safety of Denosumab in Japanese Osteoporotic Subjects With Prevalent Fragility Vertebral Fracture(s)
Brief Title: Denosumab Fracture Intervention Randomized Placebo Controlled Trial in Japanese Patients With Osteoporosis
Acronym: DIRECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMG162-A-J301
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Denosumab (subcutaneously - every 6 months) + daily calcium and vitamin D supplements for 24 months, followed by a 12-month period of denosumab (subcutaneously - every 6 months).
  Interventions: Drug: Denosumab
- 2 (Placebo Comparator): Placebo (subcutaneously every 6 months) + daily calcium and vitamin D supplements for 24 months, followed by a 12-month period of denosumab (subcutaneously - every 6 months).
  Interventions: Drug: Placebo
- 3 (Active Comparator): Alendronate sodium hydrate oral tablets weekly + daily calcium and vitamin D supplements for 24 months (open label reference arm).
  Interventions: Drug: Alendronate sodium hydrate

INTERVENTIONS:
Drug: Denosumab — Subcutaneous injection every 6 months for 24 months, followed by a 12-month period of denosumab (subcutaneously - every six months).
  Arms: 1
Drug: Placebo — Subcutaneous injection every 6 months for 24 months, followed by a 12-month period of denosumab (subcutaneously - every six months).
  Arms: 2
Drug: Alendronate sodium hydrate — Oral tablet once a week for 24 months
  Arms: 3

SUMMARY:
Evaluate the efficacy and safety of denosumab in the treatment of involutional (postmenopausal and senile) osteoporotic subjects with prevalent fragility vertebral fracture(s)

ELIGIBILITY:
Inclusion Criteria:

* Involutional (postmenopausal and senile) osteoporosis with prevalent fragility vertebral fractures

Exclusion Criteria:

* Any underlying condition,(other than BMD) that might have resulted in abnormal bone metabolism

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1262 (Actual)
Dates: Start 2008-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daiichi Sankyo, Study Chair — R&D Division, Daiichi Sankyo Co., Ltd.
Locations (4):
- Japan (4):
  - Fukuoka
  - Osaka
  - Sapporo
  - Tokyo

REFERENCES:
- [Result] Nakamura T, Matsumoto T, Sugimoto T, Hosoi T, Miki T, Gorai I, Yoshikawa H, Tanaka Y, Tanaka S, Sone T, Nakano T, Ito M, Matsui S, Yoneda T, Takami H, Watanabe K, Osakabe T, Shiraki M, Fukunaga M. Clinical Trials Express: fracture risk reduction with denosumab in Japanese postmenopausal women and men with osteoporosis: denosumab fracture intervention randomized placebo controlled trial (DIRECT). J Clin Endocrinol Metab. 2014 Jul;99(7):2599-607. doi: 10.1210/jc.2013-4175. Epub 2014 Mar 19. PMID 24646104
- [Result] Sugimoto T, Matsumoto T, Hosoi T, Miki T, Gorai I, Yoshikawa H, Tanaka Y, Tanaka S, Fukunaga M, Sone T, Nakano T, Ito M, Matsui S, Yoneda T, Takami H, Watanabe K, Osakabe T, Okubo N, Shiraki M, Nakamura T. Three-year denosumab treatment in postmenopausal Japanese women and men with osteoporosis: results from a 1-year open-label extension of the Denosumab Fracture Intervention Randomized Placebo Controlled Trial (DIRECT). Osteoporos Int. 2015 Feb;26(2):765-74. doi: 10.1007/s00198-014-2964-2. Epub 2014 Nov 18. PMID 25403903
- [Derived] Okubo N, Matsui S, Matsumoto T, Sugimoto T, Hosoi T, Osakabe T, Watanabe K, Takami H, Shiraki M, Nakamura T. Relationship Between Bone Mineral Density and Risk of Vertebral Fractures with Denosumab Treatment in Japanese Postmenopausal Women and Men with Osteoporosis. Calcif Tissue Int. 2020 Dec;107(6):559-566. doi: 10.1007/s00223-020-00750-y. Epub 2020 Aug 25. PMID 32839843

RESULTS

PARTICIPANT FLOW:
Groups:
- Denosumab: Denosumab (subcutaneously - every 6 months) + daily calcium and vitamin D supplements for 24 months, followed by a 12-month period of denosumab (subcutaneously - every 6 months).
- Placebo: Placebo (subcutaneously every 6 months) + daily calcium and vitamin D supplements for 24 months, followed by a 12-month period of denosumab (subcutaneously - every 6 months).
- Alendronate: Alendronate sodium hydrate oral tablets weekly + daily calcium and vitamin D supplements for 24 months (open label reference arm).
Period: Overall Study
Arm/Group | Denosumab | Placebo | Alendronate
Started | 500 | 511 | 251
Completed | 414 | 416 | 204
Not Completed | 86 | 95 | 47

BASELINE CHARACTERISTICS:
Population: The demography information shows the number of participants included in the full analysis set (FAS) for efficacy analyses, which includes all randomized subjects except for those who did not have osteoporosis, did not receive the investigational product, or had no available efficacy data after the first dose of the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab | Placebo | Alendronate | Total
Number analyzed (Participants) | 472 | 480 | 242 | 1194
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.36) | 69.0 (7.67) | 70.2 (7.31) | 69.6 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 449 | 456 | 230 | 1135
  Male | 23 | 24 | 12 | 59
Region of Enrollment [Number; unit: participants]
  Japan | 472 | 480 | 242 | 1194
the number of participants with vertebral fractures [Number; unit: Participants] — the number of participants with vertebral fractures
  Participants | 466 | 471 | 237 | 1174

OUTCOME MEASURES:

1. Primary Outcome: Incidence of New or Worsening Vertebral Fractures in Osteoporotic Subjects Treated With Denosumab Compared to Placebo
Time Frame: Baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: Vertebral fractures
Arm/Group | Denosumab | Placebo | Alendronate
Number analyzed (Participants) | 472 | 480 | 242
Vertebral fractures | 3.6 [2.2 to 5.8] | 10.3 [7.8 to 13.5] | 7.2 [4.6 to 11.4]
Statistical Analysis 1: Comparison: Denosumab vs Placebo; Test type: Superiority or Other; p = 0.0001, Log Rank; Hazard Ratio (HR) = 0.343, 95% CI 2-sided [0.194 to 0.606]

2. Secondary Outcome: The Percentage of Non-vertebral Fractures
Description: The results are expressed as percentage by Kaplan-Meier estimate the percentage of participants with non-vertebral fractures
Time Frame: Baseline to 24 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Denosumab | Placebo | Alendronate
Number analyzed (Participants) | 472 | 480 | 242
percentage of participants | 4.1 [2.6 to 6.6] | 4.1 [2.6 to 6.5] | 2.7 [1.2 to 5.9]
Statistical Analysis 1: Comparison: Denosumab vs Placebo; Test type: Superiority or Other; p = 0.9951, Log Rank

3. Secondary Outcome: Percentage of Participants With Hip Fractures in Osteoporotic Participants Treated With Denosumab Compared to Treatment With Placebo.
Description: The results are expressed as a percentage by Kaplan-Meier estimate.
Time Frame: Baseline to 24 Months
Measure: Number; unit: percentage of participants
Arm/Group | Denosumab | Placebo | Alendronate
Number analyzed (Participants) | 472 | 480 | 242
percentage of participants | 0.0 [0.0 to 0.0] | 0.5 [0.1 to 1.9] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Denosumab vs Placebo; Test type: Superiority or Other; p = 0.1568, Log Rank

ADVERSE EVENTS:
Time Frame: Baseline to 24 months
Description: The number of participants for which serious adverse reactions are reported are the ones included in the safety data analysis set. This data set includes all participants who received at least one dose of investigational product.
Arm/Group | Denosumab | Placebo | Alendronate
Serious Adverse Events (participants affected / at risk) | 65/475 | 68/481 | 30/242
Other Adverse Events (participants affected / at risk) | 475/475 | 481/481 | 242/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=475) | Placebo (N=481) | Alendronate (N=242)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heat illness (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 1 | 0
Cerebral infarction (Nervous system disorders) | 3 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 2 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 2 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 1
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal mucosal exfoliation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Paget's disease of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 7 | 5
Maculopathy (Eye disorders) | 1 | 1 | 1
Macular degeneration (Eye disorders) | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 1
Device dislocation (General disorders) | 1 | 0 | 0
Device breakage (General disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Dysthymic disorder (Psychiatric disorders) | 1 | 0 | 0
Neurosis (Psychiatric disorders) | 0 | 1 | 0
Cataract operation (Surgical and medical procedures) | 2 | 0 | 0
Varicose vein operation (Surgical and medical procedures) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Mixed incontinence (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 2 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal relaxation (Reproductive system and breast disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab (N=475) | Placebo (N=481) | Alendronate (N=242)
Nasopharyngitis (Infections and infestations) | 211 | 203 | 93
Cystitis (Infections and infestations) | 28 | 29 | 9
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 77 | 43 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 69 | 60 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 30 | 17
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 27 | 24 | 14
Periarthritis (Musculoskeletal and connective tissue disorders) | 23 | 26 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 25 | 12
Dental caries (Gastrointestinal disorders) | 73 | 64 | 29
Constipation (Gastrointestinal disorders) | 49 | 37 | 21
Periodontitis (Gastrointestinal disorders) | 41 | 27 | 16
Stomatitis (Gastrointestinal disorders) | 35 | 24 | 7
Diarrhoea (Gastrointestinal disorders) | 23 | 15 | 16
Gastritis (Gastrointestinal disorders) | 20 | 26 | 13
Contusion (Injury, poisoning and procedural complications) | 80 | 74 | 54
Eczema (Skin and subcutaneous tissue disorders) | 39 | 41 | 16
Dermatitis contact (Skin and subcutaneous tissue disorders) | 21 | 28 | 14
Blood creatine phosphokinase increased (Investigations) | 28 | 22 | 15
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 31 | 35 | 19
Cataract (Eye disorders) | 25 | 27 | 14
Hypertension (Vascular disorders) | 39 | 36 | 11
Insomnia (Psychiatric disorders) | 26 | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator shall not publish the results of the Study at any time without the prior written approval of Sponsor.